CLINICAL TRIAL: NCT03647293
Title: Ultrasound Guided Central Line Insertion in Neonates: Pain Score Results From a Prospective Study
Brief Title: Less Pain in Neonates During Central Lines Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint George Hospital (Other)
Responsible Party: Principal Investigator, Dany Al-Hamod, Associate Professor in Pediatrics, Head of the Post-Graduate Medical Education Office, Saint George Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB/O/036-16/1916
Record Dates: First submitted 2018-08-15; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Central Venous Catheter; Neonates; Pain
Keywords: Central Catheter; Central Line; Internal Jugular Vein; Neonate; Peripherally Inserted Central Line; Ultrasound Guided; Pain Score
MeSH Terms: conditions — Pain | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Neonates who underwent a peripherally inserted central catheter
  Interventions: Procedure: Peripherally Inserted Central Catheter
- Intervention Group (Active Comparator): Neonates who underwent an Ultrasound Guided Central Catheter Insertion
  Interventions: Procedure: Ultrasound Guided Central Catheter Insertion

INTERVENTIONS:
Procedure: Ultrasound Guided Central Catheter Insertion
  Arms: Intervention Group
Procedure: Peripherally Inserted Central Catheter
  Arms: Control Group

SUMMARY:
Central venous access is an imperative measure used in neonates whether being a peri-operative measure for children undergoing cardiac procedures for congenital heart diseases or as a mean of nutrition in neonatal enteral malnutrition and drug administration in oncology patients. Central catheters fall into two categories, a peripherally inserted central catheter (PICC) line or centrally inserted central catheters (CICC). Although these two modalities practically have the same aim, identifying the more effective technique is imperative for deciding which procedure should be applied to ameliorate patient outcomes. Many studies have been previously done that delineate the indications for central venous access with practically no absolute contraindications. These indications include central venous pressure (CVP) monitoring, poor venous access, volume resuscitation, and prolonged venous access in critically ill patients, total parenteral nutrition (TPN), cardio-pulmonary resuscitation and medication administration. Centrally inserted catheters have evolved from being blindly inserted catheters using landmarks techniques, is the usual standard of care, to being placed under direct visualization using ultrasound guidance. Since its first use back in the 90's, ultrasound guided insertion of central venous catheters has gained attention and successful attempts have been made to improve this technique. US-guidance initially used acoustic Doppler techniques but is now largely replaced by two-dimensional (2D) imaging and internal jugular vein (IJV) being the preferred site of insertion by US over femoral and subclavian vein. Several studies have compared these two techniques. Small-caliber vessels remain a great challenge in the pediatric population which backup the use of imaging modalities for a successful and safer insertion of CVCs.

This study aims to develop a better understanding of pain during central line insertions, compare pain scores between the two techniques in order to adopt the less painful technique and ultimately provide insight about the use of analgesics during these procedures for a better outcome.

DETAILED DESCRIPTION:
A single-center prospective randomized controlled study of neonates (preterm and term babies) who underwent an elective or emergent central line insertion between November 2016 and May 2017 was conducted at SGHUMC Neonatal Intensive Care Unit. Hospital's Institutional Review Board approved the study and an informed parental consent was signed for study entry. Inclusion criteria included neonates requiring TPN, antibiotic therapy for at least 7 days, and babies with poor or difficult venous access. Exclusion criteria included refusal to sign consent, patients with previously attempted or placed central lines, and patients who were converted from one technique to the other. Patients were randomized into the control and intervention group through a flip of coin each time a patient enrolled in the study The catheter used for all the patients was an epicutaneo-cava-catheter (ECC), silicone tube material kit, 24G, VYGON® (Aachen, Germany). All procedures were performed under sterile precautions such as hand washing, use of sterile gloves and gowns, facemask, hair cover, and protective eyewear.

The control group consisted of neonates who underwent a PICC line placement. The method of insertion performed followed the procedure previously described by Pettit. Patients in the intervention group underwent US-IJV. This procedure was carried out as follows: The patient's skin was sterilized with chlorhexidine gluconate and the area was infiltrated with local anesthetic agent (lidocaine). Vascular cannulation was performed using the ECC's winged needle. The target vessel was located via the US dynamic (real-time) method. At the point of needle insertion, the ECC was placed through the needle without guide wire placement. Once the catheter was inserted, a gentle aspiration was performed to show blood flow through the 3 ml syringe that was connected to the ECC. The catheter was then secured and fixed with simple steri-strips and covered by the transparent dressing. Both techniques were performed by two institutional neonatologists who according to their expertise, one performed all PICC line placements while the other performed all US-IJV.

Transducer selection and the axis of visualization are important to consider in the use of US for ECC, as such a linear 6-13 MHz transducer Sonosite M-turbo was used (manufacturer's recommendations). The transverse view shows the vessel under the transducer and the adjacent structures. The tip of the needle is visualized and inserted at a 45° angle. The longitudinal view helps to track the needle progression toward the IJV. Post procedural chest radiography was done for both groups to confirm placement and evaluate for complications.

The primary outcome measured was the pain score difference between Ultrasound inserted central line and peripherally inserted central line. The pain score was measures using the Neonatal Pain, Agitation and Sedation Scale (N -PASS). The N-PASS is based on several criteria: crying / irritability, behavior / state, facial expression, extremities / tone and vital signs. Patient characteristics such as gestational age, age, gender, admission diagnosis, weight have been taken into account and the scores was recorded by the nurse in charge of the baby before and during the procedure. Pain score difference was calculated by subtracting the score during the procedure from the pain score before the procedure.

The secondary outcome measures included the number of first successful attempts, number of total attempts and procedure duration. Additional patient information collected included gender, TPN administration, gestational age, birth weight and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* neonates requiring TPN
* antibiotic therapy for at least 7 days
* babies with poor or difficult venous access

Exclusion Criteria:

* refusal to sign consent
* patients with previously attempted or placed central lines
* patients who were converted from one technique to the other

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain score difference | Through study completion, around 7 months
  The patient pain score will be assessed prior to the procedure and during. The difference in pain score will be calculated as a representation of the increased pain inflicted by the procedure itself. This difference in pain scores will be compared across the 2 different interventions

SECONDARY OUTCOMES:
The number of first successful attempts | Through study completion, around 7 months
  With each procedure the number of attempts will be registered for each procedure, comparing between the 2 different interventions the number of successful attempts from first trial.
Number of total attempts | Through study completion, around 7 months
  With each procedure the number of attempts will be registered for each procedure, the total number of trials will be compared between the 2 different interventions
Procedure duration | Through study completion, around 7 months
  The procedure duration is the time from the start of the procedure till successful insertion of the central catheter. The total procedural duration will be compared between the 2 different interventions

CONTACTS AND LOCATIONS:
Overall Officials: Dany Al Hamod, MD, Principal Investigator — Saint Georges Hospital University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trieschmann U, Cate UT, Sreeram N. Central venous catheters in children and neonates - what is important? Images Paediatr Cardiol. 2007 Oct;9(4):1-8. PMID 22368674
- [Background] Cheung E, Baerlocher MO, Asch M, Myers A. Venous access: a practical review for 2009. Can Fam Physician. 2009 May;55(5):494-6. No abstract available. PMID 19439704
- [Background] Taylor RW, Palagiri AV. Central venous catheterization. Crit Care Med. 2007 May;35(5):1390-6. doi: 10.1097/01.CCM.0000260241.80346.1B. PMID 17414086
- [Background] Bhatt et al. Indications and complications of central venous catheterization in critically ill children in intensive care unit. National Journal of Medical Research 2012;2:1.85-88.
- [Background] Kumar A, Chuan A. Ultrasound guided vascular access: efficacy and safety. Best Pract Res Clin Anaesthesiol. 2009 Sep;23(3):299-311. doi: 10.1016/j.bpa.2009.02.006. PMID 19862889
- [Background] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Background] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Ultrasound-guided internal jugular venous cannulation in infants: a prospective comparison with the traditional palpation method. Anesthesiology. 1999 Jul;91(1):71-7. doi: 10.1097/00000542-199907000-00013. PMID 10422930
- [Background] Goldstein SD, Pryor H, Salazar JH, Dalesio N, Stewart FD, Abdullah F, Colombani P, Lukish JR. Ultrasound-Guided Percutaneous Central Venous Access in Low Birth Weight Infants: Feasibility in the Smallest of Patients. J Laparoendosc Adv Surg Tech A. 2015 Sep;25(9):767-9. doi: 10.1089/lap.2014.0308. Epub 2015 Jul 13. PMID 26168162
- [Background] Al Hamod DA, Zeidan S, Al Bizri A, Baaklini G, Nassif Y. Ultrasound-guided Central Line Insertion and Standard Peripherally Inserted Catheter Placement in Preterm Infants: Comparing Results from Prospective Study in a Single-center. N Am J Med Sci. 2016 May;8(5):205-9. doi: 10.4103/1947-2714.183011. PMID 27298814
- [Background] Pettit J. Technological advances for PICC placement and management. Adv Neonatal Care. 2007 Jun;7(3):122-31. doi: 10.1097/01.anc.0000278210.18639.fd. PMID 17844776
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn; American Academy of Pediatrics Section on Surgery; Canadian Paediatric Society Fetus and Newborn Committee; Batton DG, Barrington KJ, Wallman C. Prevention and management of pain in the neonate: an update. Pediatrics. 2006 Nov;118(5):2231-41. doi: 10.1542/peds.2006-2277. PMID 17079598
- [Background] Costa P, Camargo P, Bueno M, Kimura A. Measuring pain in neonates during placement of central line catheter via peripheral insertion. Acta Paul Enferm 2010;23(1):35-40.
- [Background] Davidson A, Flick RP. Neurodevelopmental implications of the use of sedation and analgesia in neonates. Clin Perinatol. 2013 Sep;40(3):559-73. doi: 10.1016/j.clp.2013.05.009. Epub 2013 Jul 12. PMID 23972757
- [Background] Walker SM. Neonatal pain. Paediatr Anaesth. 2014 Jan;24(1):39-48. doi: 10.1111/pan.12293. Epub 2013 Nov 13. PMID 24330444